CLINICAL TRIAL: NCT06977594
Title: A Randomized, Placebo-controlled, Parallel-group, Open-label Trial to Evaluate the Efficacy of Proactive Immune Tolerance Induction to Paclitaxel and Carboplatin in Patients With Gynecologic Cancer
Brief Title: Proactive Immune Tolerance Induction in Chemotherapy for Gynecologic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other); Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Hye-Ryun Kang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PINTO_C
Record Dates: First submitted 2025-05-03; First posted 2025-05-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Cervical Cancer
Keywords: Immune tolerance induction; Desensitization; Drug hypersensitivity; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Drug Hypersensitivity | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, parallel-group, open-label, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- (Trial 1) Proactive immune tolerance induction with 20 mg dexamethasone as premedication (Experimental): Participants will receive proactive immune tolerance induction during the first three cycles of chemotherapy, followed by standard treatment in the remaining cycles. Premedication includes 20 mg of dexamethasone.
  Interventions: Other: Proactive immune tolerance induction; Drug: Paclitaxel and carboplatin; Drug: Standard premedication (20 mg)
- (Trial 1) Standard treatment (placebo) with 20 mg dexamethasone as premedication (Active Comparator): Participants will receive standard treatment throughout all chemotherapy cycles. Premedication includes 20 mg of dexamethasone.
  Interventions: Other: Standard Treatment; Drug: Paclitaxel and carboplatin; Drug: Standard premedication (20 mg)
- (Trial 2) Proactive immune tolerance induction with 10 mg dexamethasone as premedication (Experimental): Participants will receive proactive immune tolerance induction during the first three cycles of chemotherapy, followed by standard treatment in the remaining cycles. Premedication includes 10 mg of dexamethasone.
  Interventions: Other: Proactive immune tolerance induction; Drug: Paclitaxel and carboplatin; Drug: Reduced premedication (10 mg)
- (Trial 2) Standard treatment (placebo) with 20 mg dexamethasone as premedication (Active Comparator): Participants will receive standard treatment throughout all chemotherapy cycles. Premedication includes 20 mg of dexamethasone.
  Interventions: Other: Standard Treatment; Drug: Paclitaxel and carboplatin; Drug: Standard premedication (20 mg)
- (Trial 3) Proactive immune tolerance induction with 5 mg dexamethasone as premedication (Experimental): Participants will receive proactive immune tolerance induction during the first three cycles of chemotherapy, followed by standard treatment in the remaining cycles. Premedication includes 5 mg of dexamethasone.
  Interventions: Other: Proactive immune tolerance induction; Drug: Paclitaxel and carboplatin; Drug: Reduced premedication (5 mg)
- (Trial 3) Standard treatment (placebo) with 20 mg dexamethasone as premedication (Active Comparator): Participants will receive standard treatment throughout all chemotherapy cycles. Premedication includes 20 mg of dexamethasone.
  Interventions: Other: Standard Treatment; Drug: Paclitaxel and carboplatin; Drug: Standard premedication (20 mg)

INTERVENTIONS:
Other: Proactive immune tolerance induction — Proactive immune tolerance induction during the first three cycles of chemotherapy, followed by standard treatment in the remaining cycles
  Arms: (Trial 1) Proactive immune tolerance induction with 20 mg dexamethasone as premedication; (Trial 2) Proactive immune tolerance induction with 10 mg dexamethasone as premedication; (Trial 3) Proactive immune tolerance induction with 5 mg dexamethasone as premedication
Other: Standard Treatment — Standard treatment throughout all chemotherapy cycles
  Arms: (Trial 1) Standard treatment (placebo) with 20 mg dexamethasone as premedication; (Trial 2) Standard treatment (placebo) with 20 mg dexamethasone as premedication; (Trial 3) Standard treatment (placebo) with 20 mg dexamethasone as premedication
Drug: Paclitaxel and carboplatin — A chemotherapy regimen for gynecologic cancers.
Drug: Standard premedication (20 mg) — Premedication includes 20 mg of dexamethasone.
  Arms: (Trial 1) Proactive immune tolerance induction with 20 mg dexamethasone as premedication; (Trial 1) Standard treatment (placebo) with 20 mg dexamethasone as premedication; (Trial 2) Standard treatment (placebo) with 20 mg dexamethasone as premedication; (Trial 3) Standard treatment (placebo) with 20 mg dexamethasone as premedication
Drug: Reduced premedication (10 mg) — Premedication includes 20 mg of dexamethasone.
  Arms: (Trial 2) Proactive immune tolerance induction with 10 mg dexamethasone as premedication
Drug: Reduced premedication (5 mg) — Premedication includes 5 mg of dexamethasone.
  Arms: (Trial 3) Proactive immune tolerance induction with 5 mg dexamethasone as premedication

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of proactive immune tolerance induction of chemotherapy (paclitaxel and carboplatin) for patients with gynecologic cancer.

The main questions it aims to answer are:

- Does immune tolerance induction during the first three cycles of chemotherapy reduce the incidence of hypersensitivity reactions in the remaining cycles?

Participants will:

* Undergo immune tolerance induction or standard treatment during the first three cycles of chemotherapy as randomized, after which all participants will continue the remaining cycles with standard treatment.
* Receive a reduced dose of dexamethasone premedication if assigned to the experimental group, depending on the specific protocol of each clinical trial.

DETAILED DESCRIPTION:
Proactive immune tolerance induction is applied using an automated infusion pump with a pre-programmed protocol. It follows the same stepwise dosing scheme as conventional desensitization therapy used in patients who have experienced hypersensitivity reactions before. However, it is uniquely performed in patients without a prior history of hypersensitivity reactions, aiming to prevent sensitization itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving paclitaxel and carboplatin chemotherapy for gynecologic malignancies.
* Patients with no prior history of hypersensitivity reactions to paclitaxel or carboplatin.
* Patients who are able to read and voluntarily provide written informed consent.
* Aged 19 years or older.

Exclusion Criteria:

* Patients who do not wish to participate in this study voluntarily.
* Patients who, in the opinion of the investigator, are unsuitable for participation in this clinical trial.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Hypersensitivity reaction incidence | From the initiation of each chemotherapy cycle to 2 weeks after its administration in each patient (to identify not only immediate but also delayed hypersensitivity reactions).
  Hypersensitivity reaction incidence (%) is calculated as (number of hypersensitivity reaction cases / total chemotherapy administrations) × 100.
  Hypersensitivity reaction will be defined as a Grade ≥2 event according to Common Terminology Criteria for Adverse Events (CTCAE), or a moderate or higher event according to Brown's criteria.

SECONDARY OUTCOMES:
Chemotherapy completion rate | From chemotherapy initiation to the last cycle in each patient, an average of 6 months
  Chemotherapy completion rate is defined as the proportion of patients who completed all planned chemotherapy cycles as originally scheduled at treatment initiation.
Severity of hypersensitivity reaction | From the initiation of each chemotherapy cycle to 2 weeks after its administration in each patient (to identify not only immediate but also delayed hypersensitivity reactions).
  Severity of hypersensitivity reactions will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE).
Patients' quality of life | From chemotherapy initiation to the last cycle, an average of 6 months
  Patients' quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores range from 0 to 100. Higher scores indicate better outcomes for the Global Health Status and Functional Scales, whereas higher scores on the Symptom Scales indicate worse symptoms.
Tumor Response Rate | At every third chemotherapy cycle in each patient
  Tumor response rate is defined as the proportion of patients who experience tumor size reduction or disappearance in response to chemotherapy. It is calculated as the proportion of patients who achieve a complete response (disappearance of all tumors with no evidence of new lesions) or a partial response (at least a 30% reduction in the size of tumors, with no appearance of new lesion) after planned chemotherapy.
Survival rate | At study completion in each patient, an average of 1 year
  Survival rate is defined as the proportion of patients who remain alive, with or without disease, after completion of the planned chemotherapy.
Recurrence Rate | At study completion in each patient, an average of 1 year
  Recurrence rate is defined as the proportion of patients who experience a return of disease after achieving a response to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to institutional policies regarding data confidentiality.